CLINICAL TRIAL: NCT05432713
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LP-168 Following Single and Multiple Oral Administration to Healthy Volunteers
Brief Title: A Study of LP-168 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Lupeng Pharmaceutical Company LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP-168-CN102
Record Dates: First submitted 2022-06-14; First posted 2022-06-27 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Multiple Sclerosis; NMO Spectrum Disorder
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LP-168 tablet (Experimental): After confirmation of inclusion, subjects will be randomized into the LP-168 tablet or LP-168 placebo tablet arm and receive single or multiple doses of LP-168 tablet or LP-168 placebo tablet.
  Interventions: Drug: LP-168 tablet
- LP-168 Placebo tablet (Placebo Comparator): After confirmation of inclusion, subjects will be randomized into the LP-168 tablet or LP-168 placebo tablet arm and receive single or multiple doses of LP-168 tablet or LP-168 placebo tablet.
  Interventions: Drug: LP-168 Placebo tablet

INTERVENTIONS:
Drug: LP-168 tablet — Lp-168 is a small molecule kinase inhibitor that is administered once daily via oral administration
  Other Names: NWP-775
  Arms: LP-168 tablet
Drug: LP-168 Placebo tablet — LP-168 placebo tablets contain excipients for LP-168 tablets, but do not contain the active ingredients of the drug, and are used for comparison in clinical trials with the same usage and dosage as LP-168 tablets
  Other Names: NWP-775 Placebo
  Arms: LP-168 Placebo tablet

SUMMARY:
This is a Phase I study designed to assess the safety, tolerability and pharmacokinetics of LP-168 in healthy human volunteers.

DETAILED DESCRIPTION:
This study will enroll 70 healthy subjects, will set 4 SAD and 3 MAD dose cohorts, with 10 subjects in each dose cohort. Subjects will be assigned to L-168 or placebo group by ratio of 8:2 in each cohort. Sentinel subjects will be used in each dose cohort during the single dose phase.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have no history of serious digestive system, central nervous system, cardiovascular system, kidney, respiratory system, metabolism and endocrine, skeletal and muscular system, blood system disease and cancer
* Subjects (including partners) are willing to take effective contraception measures during study and within 3 months after last dose
* Male and female healthy subjects aged 18 to 55 years old
* Male subjects weigh ≥ 50 kg, and female subjects weigh ≥ 45 kg
* Subjects able to understand and comply with study requirements
* Willing to sign the informed consent

Exclusion Criteria:

* Abnormal vital signs, physical examination or laboratory tests with clinical significance
* Abnormal ECG or echocardiography with clinical significance
* Hepatitis B virus, Hepatitis C virus, HIV and syphilis test positive. COVID-19 DNA positive.
* Subjects who have taken any drugs or health care products within 14 or 28 days before administration the study drug
* Subjects who have consumed diets that may alter the activity of liver metabolic enzymes within 7 days before administration the study drug
* Subjects who have consumed tea or alcohol-containing food product within 24hrs before administration the study drug
* Subjects who have a history of dysphagia or condition may affect drug absorption, distribution, metabolism and excretion
* Female subjects are breastfeeding or pregnant
* Subjects who have a history of drug/ alcohol/ tobacco abuse
* Subjects who have had a blood donation or massive blood loss within three months before screening; or had surgery within six months before screening
* Subjects who have participated in other clinical trial within three months before screening
* Subjects have special dietary requirements or cannot tolerate a standard meal

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-05-14 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events as determined by CTCAE v5.0 | From the first dose of the study drug to 5 days after last dose
Severity of Treatment Emergent Adverse Events as determined by CTCAE v5.0 | From the first dose of the study drug to 5 days after last dose
Pharmacokinetics (PK) As Assessed By Maximum Observed Plasma Concentration (Cmax) of LP-168 | Up to 96 hours post last dose
PK As Assessed By Area Under The Plasma Concentration Time Curve From Time 0 To The Time of The Last Quantifiable Concentration (AUC0-t) Of LP-168 | Up to 96 hours post last dose
PK As Assessed By Time To Maximum Observed Plasma Concentration (Tmax) of LP-168 | Up to 96 hours post last dose
PK As Assessed By Terminal Half-life (t1/2) of LP-168 | Up to 96 hours post last dose
PK As Assessed By Terminal Vd/F of LP-168 | Up to 96 hours post last dose
PK As Assessed By Terminal CL/F of LP-168 | Up to 96 hours post last dose

SECONDARY OUTCOMES:
PD as Assessed by elisa analysis the proportion of LP-168 occupied kinase at scheduled timepoints pre-dose and post-dose | Up to 48 hours post last dose

CONTACTS AND LOCATIONS:
Overall Officials: Jinliang Chen, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No